CLINICAL TRIAL: NCT04298216
Title: Evaluation of Transhepatic Versus Subcostal Inferior Vena Cava Views to Assess Inferior Vena Cava Variation in Pediatric Patients
Brief Title: Transhepatic Versus Subcostal Views to Assess Inferior Vena Cava Variation in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 55097
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Inferior Vena Cava Abnormality

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Assessment of Inferior Vena Cavae with Subcostal View (Active Comparator): Patients will have a novel operator attempt to visualize their Inferior Vena Cavae with the probe placed in the subcostal region.
  Interventions: Diagnostic Test: Ultrasound Analysis of Inferior Vena Cavae (IVC)
- Assessment of Inferior Vena Cavae with Transhepatic View (Experimental): Patients will have a novel operator attempt to visualize their Inferior Vena Cavae with the probe placed in the transhepatic region.
  Interventions: Diagnostic Test: Ultrasound Analysis of Inferior Vena Cavae (IVC)

INTERVENTIONS:
Diagnostic Test: Ultrasound Analysis of Inferior Vena Cavae (IVC) — Novel Operators will attempt to visualize the Inferior Vena Cavae through two different views on the patient's body. The images taken will be interpreted by an expert ultrasound user to determine if the novel operator was successful in locating and evaluating the IVC.

SUMMARY:
Currently, in order to visualize the inferior vena cava (IVC) of the heart using ultrasound, physicians traditionally place the ultrasound probe onto the "Subcostal" area which is located below the chest in the upper abdomen area. In this location, the pressure from the ultrasound probe is often uncomfortable for adults, and even more so for pediatric patients. Previous research and physician experience have demonstrated that it is possible to visualize the heart in the "transhepatic" area which is located under the arm on the side of the chest. By placing the ultrasound probe in this location, it is more comfortable for the patient when applying pressure, and this study aims to prove the effectiveness of visualizing the heart through this new location.

ELIGIBILITY:
Inclusion Criteria:

1. Be between ages of 2-18 years of age
2. Have parental consent
3. located at an inpatient/outpatient facility at LPCH
4. Be hemodynamically stable

Exclusion Criteria:

1. Emergent Surgical Procedures
2. BMI greater than 24

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Time | For the entirety of the ultrasound procedure.
  Novel Operators will be timed from the point at which the probe is placed until the image has been and will be evaluated between both the control and experimental groups.
Accuracy of the IVC Analysis | For the entirety of the ultrasound procedure.
  Novel Operators will be evaluated by the ultrasound expert who will confirm clinical success in locating the IVC.

IPD SHARING:
Plan to Share IPD: No